CLINICAL TRIAL: NCT02585960
Title: Phase 3, Prospective, Randomized, Multi-center Clinical Study Comparing the Safety and Efficacy of BAX 855 Following PK-guided Prophylaxis Targeting Two Different FVIII Trough Levels in Subjects With Severe Hemophilia A
Brief Title: BAX 855 PK-guided Dosing
Acronym: PROPEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 261303; 2014-005477-37 (EudraCT Number)
Record Dates: First submitted 2015-10-21; First posted 2015-10-26 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BAX 855

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pharmacokinetic (PK) evaluation of BAX 855 (Experimental): Participants will first undergo an initial pharmacokinetic (PK) assessment. Following the PK assessment participants will be randomized to one of 2 dosing regimens.
  Interventions: Biological: PEGylated Recombinant Factor VIII
- FVIII trough target 1-3% (Experimental): Standard treatment arm - PK-guided dosing schedule to achieve a Factor VIII (FVIII) trough of 1-3%
  Interventions: Biological: PEGylated Recombinant Factor VIII
- FVIII trough target 8-12% (Experimental): Intensified treatment arm - PK-guided dosing schedule to achieve a Factor VIII (FVIII) trough of 8-12%
  Interventions: Biological: PEGylated Recombinant Factor VIII

INTERVENTIONS:
Biological: PEGylated Recombinant Factor VIII — Pharmacokinetic (PK) evaluation
  Other Names: BAX855; BAX 855
  Arms: Pharmacokinetic (PK) evaluation of BAX 855
Biological: PEGylated Recombinant Factor VIII — Standard treatment
  Other Names: BAX 855; BAX855
  Arms: FVIII trough target 1-3%
Biological: PEGylated Recombinant Factor VIII — Intensified treatment
  Other Names: BAX855; BAX 855
  Arms: FVIII trough target 8-12%

SUMMARY:
1. To compare the efficacy and safety of pharmacokinetic (PK)-guided treatment with BAX 855 targeting FVIII trough levels of 1-3% and approximately 10% (8-12%)
2. To further characterize pharmacokinetic (PK) and pharmacodynamic (PD) parameters of BAX 855

ELIGIBILITY:
INCLUSION CRITERIA:

* Participants transitioning from another BAX 855 study who meet ALL of the following criteria are eligible for this study:

  1. Participant has completed the end of study visit of a BAX 855 study or is transitioning from the ongoing Baxalta Continuation Study 261302.
  2. Participant is either receiving on-demand treatment or prophylactic treatment with BAX 855 and had an Annual Bleed Rate (ABR) of ≥ 2 documented and treated during the past 12 months.
  3. Participant is human immunodeficiency virus negative (HIV-); or HIV+ with stable disease and CD4+ count ≥ 200 cells/mm^3, as confirmed by central laboratory.
  4. Participant is willing and able to comply with the requirements of the protocol.
* Newly recruited participants (ie not transitioning from another BAX 855 study) including BAX855 naïve participants who meet ALL of the following criteria are eligible for this study:

  1. Participant has severe hemophilia A (FVIII clotting activity < 1%) as confirmed by central laboratory OR by historically documented FVIII clotting activity performed by a certified clinical laboratory, optionally supported by a FVIII gene mutation consistent with severe hemophilia A
  2. Participant has been previously treated with plasma-derived FVIII concentrates or recombinant FVIII for ≥ 150 documented exposure days (EDs)
  3. Participant is either receiving on-demand treatment or prophylactic treatment and had an annual bleeding rate of ≥ 2 documented and treated during the past 12 months.
  4. Participant has a Karnofsky performance score of ≥ 60 at screening
  5. Participant is HIV-; or HIV+ with stable disease and CD4+ count ≥ 200 cells/mm^3, as confirmed by central laboratory at screening
  6. Participant is hepatitis C virus negative (HCV-) by antibody (if positive, additional PCR testing will be performed), as confirmed by central laboratory at screening; or HCV+ with chronic stable hepatitis
  7. If female of childbearing potential, participant presents with a negative urine pregnancy test and agrees to employ adequate birth control measures for the duration of the study
  8. Participant is willing and able to comply with the requirements of the protocol.

EXCLUSION CRITERIA:

* Participants transitioning from another BAX 855 study who meet ANY of the following criteria are not eligible for this study:

  1. Participant has developed a confirmed inhibitory antibody to FVIII with a titer of ≥ 0.6 BU using the Nijmegen modification of the Bethesda assay as determined at the central laboratory during the course of the previous BAX 855 study.
  2. Participant has been diagnosed with an acquired hemostatic defect other than hemophilia A.
  3. The participant's weight is < 35 kg or > 100 kg.
  4. Participant's platelet count is < 100,000/mL.
  5. Participant has an abnormal renal function (serum creatinine > 1.5 times the upper limit of normal).
  6. Participant has active hepatic disease with alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels ≥ 5 times the upper limit of normal.
  7. Participant is scheduled to receive a systemic immunomodulating drug (e.g. corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day, or α-interferon) other than anti-retroviral chemotherapy during the study.
  8. Participant has a clinically significant medical, psychiatric, or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect participant's safety or compliance.
  9. Participant is planning to take part in any other clinical study during the course of the study.
  10. Participant is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study.

Newly recruited participants (ie not transitioning from another BAX 855 study) who meet ANY of the following criteria are not eligible for this study:

1. Participant has detectable FVIII inhibitory antibodies (≥ 0.6 BU using the Nijmegen modification of the Bethesda assay) as confirmed by central laboratory at screening.
2. Participant has a history of confirmed FVIII inhibitors with a titer ≥ 0.6 Bethesda Units (BU) (as determined by the Nijmegen modification of the Bethesda assay or the assay employed with the respective cut-off in the local laboratory) at any time prior to screening.
3. Participant has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (eg, qualitative platelet defect or von Willebrand's disease).
4. The participant's weight is < 35 kg or > 100 kg.
5. Participant's platelet count is < 100,000/mL.
6. Participant has known hypersensitivity towards mouse or hamster proteins, PEG or Tween 80.
7. Participant has severe chronic hepatic dysfunction [eg, ≥ 5 times upper limit of normal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), as confirmed by central laboratory at screening, or a documented INR > 1.5].
8. Participant has severe renal impairment (serum creatinine > 1.5 times the upper limit of normal).
9. Participant has current or recent (< 30 days) use of other pegylated drugs prior to study participation or is scheduled to use such drugs during study participation.
10. Participant is scheduled to receive during the course of the study, a systemic immunomodulating drug (e.g. corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day, or α-interferon) other than anti-retroviral chemotherapy.
11. Participant has participated in another clinical study involving an IP or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
12. Participant has a medical, psychiatric, or cognitive illness or recreational drug/alcohol use that, in the opinion of the investigator, would affect participant safety or compliance.
13. Participant is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2018-08-05 (Actual); Study Completion 2018-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (83):
- United States (14):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arizona Hemophilia & Thrombosis Center, located within The University of Arizona Cancer Center, Tucson, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - Emory University-ECC, Atlanta, Georgia
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville KCPCRU, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Gulf States Hemophilia Centre, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- Australia (2):
  - Royal Brisbane Women's Hospital, Herston, Queensland
  - The Perth Blood Institute, Nedlands, Western Australia
- AKH - Medizinische Universität Wien, Vienna, Austria
- Bulgaria (3):
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - MHAT 'Sv. Marina', EAD, Clinic of Clinical Hematology, Varna
- France (5):
  - CHU Nice- Service hematologie, Nice, Alpes Maritimes
  - Hôpital Morvan, Brest, Finistere
  - CHU Rennes - Hopital Pontchaillou, Rennes, Ille Et Vilaine
  - CHU de Caen - Hôpital Côte de Nacre, Caen
  - CHU Charles Nicolle, Rouen
- Germany (5):
  - HZRM Hamophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf, Hesse
  - Inst. f. Experimentelle Hamatologie u. Transfusionsmedizin, Bonn, North Rhine-Westphalia
  - COAGULATION RESEARCH CENTRE GmbH, Duisburg, North Rhine-Westphalia
  - Hamophiliezentrum/Gerinnungssprechstunde, Berlin
  - MVZ Labor Dr. Reising-Ackermann, Leipzig
- Hong Kong (2):
  - University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Shatin
- Hungary (3):
  - Magyar Honvedseg EK, Budapest
  - DE OEC Belgyógyászati Int, Debrecen
  - PTE ÁOK, Pécs
- Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Italy (7):
  - UOC Ematologia, Azienda ULSS 8 Asolo, Regione Veneto, Castelfranco Veneto, Treviso
  - Presidio Osped. Ferrarotto, Catania
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Roma
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - AOU Citta della Salute e della Scienza - Presidio Molinette, Torino
  - ULSS n. 6 "Vicenza", Vicenza
- Malaysia (5):
  - Hospital Ampang, Ampang, Kuala Lumpur
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Melaka, Malacca
  - Hospital Pulau Pinang, Pulau Pinang
- Oslo Universitetssykehus HF, Oslo, Norway
- Poland (4):
  - Wojewodzki Szpital Specjalistyczny im. Mikolaja Kopernika, Klinika Hematologii, Lodz
  - Alvamed, Poznan
  - Instytut Hematologii Ii Transfuzjologii, Warsaw
  - SP Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw
- Romania (2):
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - Institutul Oncologic ClNa., Cluj-Napoca
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital- Parent, Singapore
  - KK Women's And Children's Hospital, Singapore
- Spain (4):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Regional Universitario de Malaga, Málaga, Málaga
  - Hospital Universitario La Paz, Madrid
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset, Stockholm
- Universitätsspital Zürich, Zurich, Switzerland
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Tri-Service General Hospital, Taipei
- Turkey (Türkiye) (4):
  - Acibadem Hastanesi, Adana
  - Akdeniz University, Antalya
  - Istanbul University, Istanbul
  - Ege University, Izmir
- Ukraine (4):
  - NChSH Okhmatdyt of MoHU Center of Children Oncohematology and Bone Marrow Transplantation, Kyiv
  - Kyiv CCH #9 Dept of Surgery City SPC of Diagnostics & Treatment of Patients with HP, Kyiv
  - SI Institute of Blood Pathology and Transfusion Medicine of NAMSU, Lviv
  - M.V. Sklifosovskyi Poltava RCH Dept of Gematology HSEIU Ukrainian Medical Stomatological Academy, Poltava
- United Kingdom (7):
  - Bristol Royal Hospital for Children, Bristol, Avon
  - Royal Free Hospital, London, Greater London
  - Royal Manchester Children's Hospital, Manchester, Greater Manchester
  - Southampton General Hospital, Southampton, Hampshire
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Churchill Hospital, Oxford, Oxfordshire
  - University Hospital of Wales, Cardiff, West Glamorgan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Escuriola-Ettingshausen C, Klamroth R, Escobar M, Stasyshyn O, Tangada S, Engl W, Honauer I, Lee HY, Chowdary P, Windyga J. Targeting an elevated FVIII level using personalized rurioctocog alfa pegol prophylaxis in specific patient populations with hemophilia A: post hoc subanalysis of the randomized, phase 3 PROPEL study. Ther Adv Hematol. 2023 Jul 15;14:20406207231178596. doi: 10.1177/20406207231178596. eCollection 2023. PMID 37465396
- [Derived] Sun SX, Crawford S. Microsimulation to compare activity-related bleed risks between pharmacokinetic-guided rurioctocog alfa pegol prophylaxis and emicizumab. Expert Rev Hematol. 2023 Mar;16(3):205-211. doi: 10.1080/17474086.2023.2162498. Epub 2023 Jan 18. PMID 36655343
- [Derived] Klamroth R, Windyga J, Radulescu V, Collins PW, Stasyshyn O, Ibrahim HM, Engl W, Tangada SD, Savage W, Ewenstein B. Rurioctocog alfa pegol PK-guided prophylaxis in hemophilia A: results from the phase 3 PROPEL study. Blood. 2021 Apr 1;137(13):1818-1827. doi: 10.1182/blood.2020005673. PMID 33150384

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 62 study centers in 19 countries between 23 November 2015 (first participant first visit) and 05 August 2018 (last participant last visit).
Pre-assignment Details: A total of 135 participants were enrolled in the study. Of them,14 participants were dropped out and did not receive any treatment 121 participants underwent initial pharmacokinetic(PK) assessment with a single administration of BAX 855 and based on their individual PK values, 115 participants were randomized to any one of the prophylactic regimen.
Groups:
- BAX 855-Low Level: Participants with severe hemophilia A received a single BAX 855 dose of 60 +/- 5 international units per kilogram (IU/kg) intravenous (IV) infusion (PK assessment) followed by a PK-guided dose of BAX 855 twice weekly (Alternating 3 and 4-day infusion intervals or an infusion every 3.5 days), targeting factor VIII (FVIII) trough levels of 1-3%. Depending on participant's individual PK, more frequent dosing was considered if single doses of greater than (>) 80 IU/kg were required or regular FVIII peak levels of 200% were reached.
- BAX 855-High Level: Participants with severe hemophilia A received a single BAX 855 dose of 60 +/- 5 IU/kg IV infusion (PK assessment) followed by a PK-guided dose of BAX 855 every other day, targeting FVIII trough levels of 8-12%. Depending on participant's individual PK, a different dosing interval was considered to prevent regular high FVIII peak levels.
- BAX 855-Non-randomized: Participants with severe hemophilia A received a single BAX 855 dose of 60 +/- 5 IU/kg IV infusion (PK assessment) and were not randomized to any treatments.
Period: PK/Safety Assessment Period
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Started | 57 | 58 | 6
Completed 1st 6 Month Period | 57 | 53 | 0
Completed 2nd 6 Month Period | 52 | 48 | 0
Completed | 52 | 48 | 0
Not Completed | 5 | 10 | 6
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 5
Not completed — Non-compliance to study procedures | 0 | 2 | 0
Not completed — Other | 4 | 4 | 0
Not completed — Withdrawn by sponsor | 0 | 1 | 0
Not completed — Screen Failure | 0 | 0 | 1
Period: Prophylactic Treatment Period
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Started | 52 | 48 | 0
Completed | 52 | 43 | 0
Not Completed | 0 | 5 | 0
Not completed — Major protocol deviation | 0 | 4 | 0
Not completed — Subject less than 75% exposed to BAX 855 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all participants enrolled who had at least one BAX 855 infusion.
Groups:
- BAX 855-Low Level: Participants with severe hemophilia A received a single BAX 855 dose of 60 +/- 5 IU/kg IV infusion (PK assessment) followed by a PK-guided dose of BAX 855 twice weekly (Alternating 3 and 4-day infusion intervals or an infusion every 3.5 days), targeting FVIII trough levels of 1-3%. Depending on participant's individual PK, more frequent dosing was considered if single doses of > 80 IU/kg were required or regular FVIII peak levels of 200% were reached.
- Total: Total of all reporting groups
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized | Total
Number analyzed (Participants) | 57 | 58 | 6 | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of informed consent was reported.
  Years | 31.1 (13.76) | 31.2 (12.22) | 25.8 (10.03) | 30.9 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 57 | 58 | 6 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 2 | 9
  Not Hispanic or Latino | 53 | 53 | 4 | 110
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 14 | 18 | 2 | 34
  White | 40 | 36 | 4 | 80
  Native Latin American | 1 | 1 | 0 | 2
  Mestizo | 0 | 1 | 0 | 1
  Other | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Total Annualized Bleeding Rate (ABR) of Zero for Second Six Months
Description: Annualized bleeding rate was determined by dividing the number of bleeds by observation period in years.
Time Frame: Day 183 to Day 364 (6 months)
Population: Full analysis set (FAS) included all participants who were randomized to one of the two prophylactic arms and treated prophylactically for any period of time.
Measure: Number; unit: Percentage of participants
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 57 | 58
Percentage of participants | 42.1 | 62.1
Statistical Analysis 1: Comparison: BAX 855-Low Level vs BAX 855-High Level; The proportion of participants with an ABR of 0 during the second 6-month period on BAX 855 prophylaxis, was compared between the 2 prophylaxis arms using a chi-square test with continuity correction at a 2-sided 5% level of significance; Test type: Superiority; p = 0.0545, Chi-squared; Gaussian Statistic estimate = 1.960, 95% CI 2-sided [-0.038 to 3.958] — Approximately Gaussian Statistic is obtained by taking the square root of the Chi-squared test with continuity adjustment

2. Secondary Outcome: Total Annualized Bleeding Rate for Second Six Months
Description: Annualized bleeding rate was determined by dividing the number of bleeds by observation period in years.
Time Frame: Day 183 to Day 364 (6 months)
Population: FAS included all participants who were randomized to one of the two prophylactic arms and treated prophylactically for any period of time. Here "Number of participants analyzed" refer to number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 57 | 53
Bleeds per year | 3.603 (7.512) | 1.649 (3.433)

3. Secondary Outcome: Annualized Spontaneous Bleeding Rate for Second Six Months
Description: Annualized spontaneous bleeding rate was determined by dividing the number of spontaneous bleeds by observation period in years. A bleed was defined as spontaneous if it was not related to injury/trauma.
Time Frame: Day 183 to Day 364 (6 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Bleeds per year
Groups:
- BAX 855 - Low Level: Participants with severe hemophilia A received a single BAX 855 dose of 60 +/- 5 IU/kg IV infusion (PK assessment) followed by a PK-guided dose of BAX 855 twice weekly (Alternating 3 and 4-day infusion intervals or an infusion every 3.5 days), targeting FVIII trough levels of 1-3%. Depending on participant's individual PK, more frequent dosing was considered if single doses of > 80 IU/kg were required or regular FVIII peak levels of 200% were reached.
- BAX 855 - High Level: Participants with severe hemophilia A received a single BAX 855 dose of 60 +/- 5 IU/kg IV infusion (PK assessment) followed by a PK-guided dose of BAX 855 every other day, targeting FVIII trough levels of 8-12%. Depending on participant's individual PK, a different dosing interval was considered to prevent regular high FVIII peak levels.
Arm/Group | BAX 855 - Low Level | BAX 855 - High Level
Number analyzed (Participants) | 57 | 53
Bleeds per year | 2.489 (6.554) | 0.737 (1.738)

4. Secondary Outcome: Annualized Traumatic Bleeding Rate for Second Six Months
Description: Annualized traumatic bleeding rate was determined by dividing the number of traumatic bleeds by observation period in years. A bleed was defined as traumatic if it was related to injury/trauma.
Time Frame: Day 183 to Day 364 (6 months)
Population: FAS included all participants who were randomized to one of the two prophylactic arms and treated prophylactically for any period of time. Here "Number of participants analyzed" refer to number of participants evaluable for this outcome at specified time points.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 57 | 53
Bleeds per year | 1.114 (2.037) | 0.912 (2.647)

5. Secondary Outcome: Annualized Joint Bleeding Rate (AJBR) for Second Six Months
Description: Annualized joint bleeding rate was determined by dividing the number of joint bleeds by observation period in years. An acute joint bleed include some or all of the following: 'aura', pain, swelling, warmth of the skin over the joint, decreased range of motion and difficulty in using the limb compared with baseline or loss of function.
Time Frame: Day 183 to Day 364 (6 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 57 | 53
Bleeds per year | 2.617 (7.361) | 1.079 (2.553)

6. Secondary Outcome: Total Weight-adjusted Consumption of BAX 855
Description: Total weight-adjusted consumption of BAX 855 were reported.
Time Frame: From start of study treatment up to 12 months (completion or termination)
Population: FAS included all participants who were randomized to one of the two prophylactic arms and treated prophylactically for any period of time.
Measure: Mean (Standard Deviation); unit: International units per kilogram (IU/kg)
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 57 | 58
International units per kilogram (IU/kg) | 3984.593 (1678.461) | 7030.714 (3208.049)

7. Secondary Outcome: Number of Bleeding Episodes: Overall Hemostatic Efficacy Rating at Number of Infusions
Description: The participant or caregiver rated the overall treatment response using a 4-point efficacy rating scale as Excellent: Full relief of pain and cessation of objective signs of bleeding after a single infusion and no additional infusion is required for the control of bleeding; Good: Definite pain relief and/or improvement in signs of bleeding after a single infusion and possibly requires more than 1 infusion for complete resolution; Fair: Probable and/or slight relief of pain and slight improvement in signs of bleeding after a single infusion and required more than 1 infusion for complete resolution and None: No improvement or condition worsens.
Time Frame: 8 hours after study drug administration
Population: as for outcome 4
Measure: Number; unit: Treated Bleeds
Units Other Than Participants: Bleeds
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 28 | 19
Number analyzed (Bleeds) | 97 | 46
Treated Bleeds
  Excellent: Bleeds treated with 1 infusion: number analyzed (Bleeds) | 58 | 33
  Excellent: Bleeds treated with 1 infusion | 19 | 17
  Excellent: Bleeds treated with 2 infusions: number analyzed (Bleeds) | 27 | 7
  Excellent: Bleeds treated with 2 infusions | 3 | 1
  Excellent: Bleeds treated with 3 infusions: number analyzed (Bleeds) | 9 | 3
  Excellent: Bleeds treated with 3 infusions | 0 | 1
  Excellent: Bleeds treated with >= 4 infusions: number analyzed (Bleeds) | 3 | 3
  Excellent: Bleeds treated with >= 4 infusions | 0 | 0
  Good: Bleeds treated with 1 infusion: number analyzed (Bleeds) | 58 | 33
  Good: Bleeds treated with 1 infusion | 36 | 16
  Good: Bleeds treated with 2 infusions: number analyzed (Bleeds) | 27 | 7
  Good: Bleeds treated with 2 infusions | 16 | 6
  Good: Bleeds treated with 3 infusions: number analyzed (Bleeds) | 9 | 3
  Good: Bleeds treated with 3 infusions | 5 | 1
  Good: Bleeds treated with >= 4 infusion: number analyzed (Bleeds) | 3 | 3
  Good: Bleeds treated with >= 4 infusion | 2 | 2
  Fair: Bleeds treated with 1 infusion: number analyzed (Bleeds) | 58 | 33
  Fair: Bleeds treated with 1 infusion | 2 | 0
  Fair: Bleeds treated with 2 infusions: number analyzed (Bleeds) | 27 | 7
  Fair: Bleeds treated with 2 infusions | 7 | 0
  Fair: Bleeds treated with 3 infusions: number analyzed (Bleeds) | 9 | 3
  Fair: Bleeds treated with 3 infusions | 4 | 0
  Fair: Bleeds treated with >= 4 infusions: number analyzed (Bleeds) | 3 | 3
  Fair: Bleeds treated with >= 4 infusions | 1 | 0
  None: Bleeds treated with 1 infusion: number analyzed (Bleeds) | 58 | 33
  None: Bleeds treated with 1 infusion | 1 | 0
  None: Bleeds treated with 2 infusions: number analyzed (Bleeds) | 27 | 7
  None: Bleeds treated with 2 infusions | 1 | 0
  None: Bleeds treated with 3 infusions: number analyzed (Bleeds) | 9 | 3
  None: Bleeds treated with 3 infusions | 0 | 1
  None: Bleeds treated with >= 4 infusions: number analyzed (Bleeds) | 3 | 3
  None: Bleeds treated with >= 4 infusions | 0 | 1

8. Secondary Outcome: Number of Bleeding Episodes: Overall Hemostatic Efficacy Rating at Bleed Resolution
Description: as for outcome 7
Time Frame: From start of study treatment up to bleed resolution (up to 12 months)
Population: as for outcome 4
Measure: Number; unit: Treated Bleeds
Units Other Than Participants: Bleeds
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 39 | 26
Number analyzed (Bleeds) | 148 | 78
Treated Bleeds
  Excellent: Bleeds treated with 1 infusion: number analyzed (Bleeds) | 100 | 58
  Excellent: Bleeds treated with 1 infusion | 50 | 34
  Excellent: Bleeds treated with 2 infusions: number analyzed (Bleeds) | 29 | 10
  Excellent: Bleeds treated with 2 infusions | 4 | 2
  Good:Bleeds treated with 1 infusion: number analyzed (Bleeds) | 100 | 58
  Good:Bleeds treated with 1 infusion | 47 | 24
  Good:Bleeds treated with 2 infusions: number analyzed (Bleeds) | 29 | 10
  Good:Bleeds treated with 2 infusions | 19 | 7
  Good:Bleeds treated with 3 infusions: number analyzed (Bleeds) | 13 | 4
  Good:Bleeds treated with 3 infusions | 6 | 3
  Good:Bleeds treated with >= 4 infusions: number analyzed (Bleeds) | 6 | 6
  Good:Bleeds treated with >= 4 infusions | 3 | 6
  Fair:Bleeds treated with 1 infusion: number analyzed (Bleeds) | 100 | 58
  Fair:Bleeds treated with 1 infusion | 3 | 0
  Fair:Bleeds treated with 2 infusions: number analyzed (Bleeds) | 29 | 10
  Fair:Bleeds treated with 2 infusions | 5 | 1
  Fair:Bleeds treated with 3 infusions: number analyzed (Bleeds) | 13 | 4
  Fair:Bleeds treated with 3 infusions | 7 | 0
  Fair:Bleeds treated with >= 4 infusions: number analyzed (Bleeds) | 6 | 6
  Fair:Bleeds treated with >= 4 infusions | 3 | 0
  None:Bleeds treated with 2 infusions: number analyzed (Bleeds) | 29 | 10
  None:Bleeds treated with 2 infusions | 1 | 0
  None:Bleeds treated with 3 infusions: number analyzed (Bleeds) | 13 | 4
  None:Bleeds treated with 3 infusions | 0 | 1

9. Secondary Outcome: Treatment of Bleeding Episodes: Number of BAX 855 Infusions Per Bleeding Episode Required Until Bleed Resolution
Description: Infusions of BAX 855 that were required until bleed resolution were reported.
Time Frame: From start of study treatment up to 12 months (completion or termination)
Population: FAS included all participants who were randomized to one of the two prophylactic arms and treated prophylactically for any period of time. Here "Number of participants analyzed" refer to number of participants with treated bleeds.
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 41 | 26
Infusions | 1.6 (1.19) | 1.6 (1.36)

10. Secondary Outcome: Change From Baseline in Hemophilia Joint Health Score (HJHS)- Total Score
Description: HJHS was assessed based on the following components of the elbow, knee, and ankle joints: swelling, duration of swelling, muscle atrophy, crepitus on motion, flexion loss, extension loss, joint pain, and strength, together with an assessment of the global gait. The HJHS is a validated 11-item scoring tool based on radiologic and clinical evaluation, sensitive to detect early signs and minor changes. HJHS ranges from 0 to 124. Higher values in the HJHS represent worse situation for the participant.
Time Frame: Baseline, Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 57 | 54
Score on a scale | -1.9 (5.25) | -1.1 (7.77)

11. Secondary Outcome: Number of Participants With Hemostatic Efficacy Ratings for BAX 855 Treatment of Operative Bleeds
Description: The participant or caregiver rated the overall treatment response using a 4-point efficacy rating scale as Excellent: Full relief of pain and cessation of objective signs of bleeding after a single infusion and no additional infusion is required for the control of bleeding; Good: Definite pain relief and/or improvement in signs of bleeding after a single infusion and possibly requires more than 1 infusion for complete resolution; Fair: Probable and/or slight relief of pain and slight improvement in signs of bleeding after a single infusion and required more than 1 infusion for complete resolution and None: No improvement or condition worsens. Hemostatic efficacy was evaluated intra-operatively (from start to end of the procedure), post-operatively (from the end of procedure up to 24 h post procedure), and perioperatively (from the start of procedure to participant discharge from hospital or 14 days after completion of procedure; whichever was first).
Time Frame: Day 0 through discharge or 14 days post-surgery
Population: Surgery analysis set included all participants in the FAS (randomized to one of the two prophylactic arms and treated prophylactically for any period of time) who underwent some form of surgery (including dental) during the course of study participation.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 3 | 4
Participants
  Excellent: Intra-operative | 1 | 3
  Excellent: Post-operative | 3 | 4
  Excellent: Peri-operative | 2 | 4
  Good: Intra-operative | 0 | 0
  Good: Post-operative | 0 | 0
  Good: Peri-operative | 0 | 0
  Fair: Intra-operative | 0 | 1
  Fair: Post-operative | 0 | 0
  Fair: Peri-operative | 0 | 0
  None: Intra-operative | 0 | 0
  None: Post-operative | 0 | 0
  None: Peri-operative | 0 | 0
  Unknown: Intra-operative | 2 | 0
  Unknown: Post-operative | 0 | 0
  Unknown: Peri-operative | 1 | 0

12. Secondary Outcome: Blood Loss Per Participant in Case of Surgery
Description: The intraoperative blood loss was measured by determining the volume of blood and fluid removal through suction into the collection container (waste box and/or cell saver) and the estimated blood loss into swabs and towels during the procedure, per the anesthesiologist's record. Postoperatively, blood loss was determined by the drainage volume collected, which mainly consisted of drainage fluid via vacuum or gravity drain, as applicable. In cases where no drain was present, blood loss was determined by the surgeon's clinical judgment, as applicable or entered as "not available". Blood loss was evaluated intra-operatively (from start to end of the procedure), post-operatively (from the end of procedure up to 24 h post procedure), and perioperatively (from the start of procedure to participant discharge from hospital or 14 days after completion of procedure; whichever was first).
Time Frame: Day 0 through discharge or 14 days post-surgery
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 3 | 4
Milliliters (mL)
  Intra-operative: Observed | 4.400 (4.017) | 72.000 (160.741)
  Intra-operative: Predicted Average | 10.600 (9.227) | 65.833 (139.290)
  Intra-operative: Predicted Maximum | 20.800 (18.089) | 128.333 (231.790)
  Post-operative: Observed: number analyzed (Participants) | 0 | 1
  Post-operative: Observed |  | 820.000 (NA) — Standard Deviation is not calculated due to a single participant being evaluable.
  Post-operative: Predicted Average | 10.000 (9.129) | 145.000 (320.967)
  Post-operative: Predicted Maximum | 20.200 (17.987) | 230.000 (475.563)

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any unfavorable and unintended sign (an abnormal laboratory finding), symptom (rash, pain, discomfort, fever, dizziness, etc.), disease (peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an investigational product (IP), whether or not considered causally related to the IP. A SAE was defined as an untoward medical occurrence that at any dose met one or more of the following criteria: outcome was fatal/results in death, life-threatening, required in-patient hospitalization or resulted in prolongation of an existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event that was not immediately life-threatening or resulted in death or required hospitalization but jeopardize the participant or required medical or surgical intervention to prevent any of the above outcomes.
Time Frame: From start of study treatment up to 12 months (completion or termination)
Population: SAS included all participants enrolled who had at least one BAX 855 infusion.
Measure: Count of Participants; unit: Participants
Groups:
- BAX 855-Low Level: Participants with severe hemophilia A received a single BAX 855 dose of 60 +/- 5 international units per kilogram (IU/kg) intravenous (IV) infusion (PK assessment) followed by a PK-guided dose of BAX 855 twice weekly (Alternating 3 and 4-day infusion intervals or an infusion every 3.5 days), targeting FVIII trough levels of 1-3%. Depending on participant's individual PK, more frequent dosing was considered if single doses of >80 IU/kg were required or regular FVIII peak levels of 200% were reached.
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 57 | 58 | 6
Participants
  Number of Participants with SAE | 5 | 5 | 0
  Number of Participants with AE | 35 | 38 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Reported as Treatment Related Adverse Events
Description: Vital signs included systolic and diastolic blood pressure, pulse rate, respiratory rate, body temperature.
Time Frame: From start of study treatment up to 12 months (completion or termination)
Population: SAS included all participants enrolled who had at least one BAX 855 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 57 | 58 | 6
Participants | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters Reported as Treatment Related Adverse Events
Description: Clinical laboratory assessments included clinical chemistry, hematology, lipid panel, genetics, T-cell, B-cell and NK cell (TBNK) and viral serology.
Time Frame: From start of study treatment up to 12 months (completion or termination)
Population: SAS included all participants enrolled who had at least one BAX 855 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 57 | 58 | 6
Participants | 2 | 1 | 0

16. Secondary Outcome: Number of Participants With Positive Inhibitory Antibodies and Binding Antibodies to Factor VIII (FVIII), BAX 855, Polyethylene Glycol (PEG), and Chinese Hamster Ovary (CHO) Protein
Description: Positive Inhibitory Antibodies and Binding Antibodies to Factor VIII (FVIII), BAX 855, Polyethylene Glycol (PEG), and Chinese Hamster Ovary (CHO) Protein were reported here.
Time Frame: From start of study treatment up to 12 months (completion or termination)
Population: SAS included all participants enrolled who had at least one BAX 855 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 57 | 58
Participants
  Binding IgG antibodies to FVIII | 0 | 3
  Binding IgM antibodies to FVIII | 0 | 0
  Binding IgG antibodies to PEG-FVIII | 2 | 7
  Binding IgM antibodies to PEG-FVIII | 0 | 1
  Binding IgG antibodies to PEG | 0 | 0
  Binding IgM antibodies to PEG | 1 | 3
  Binding Ig antibodies to CHO | 0 | 0
  Inhibitory antibodies to FVIII | 0 | 1

17. Secondary Outcome: Change From Baseline in Physical Component Scores (PCS) of the Short Form-36 (SF-36) Health Survey
Description: Short Form (36) Health Survey (SF-36) is a 36-item validated, generic health related quality of life (HR QoL) instrument. PCS is a summary scale of the dimensions physical functioning, role physical, bodily pain, and general health. The component score is normalized to a standard population. Scores range from 0 to 100 with higher scores representing better health. There is no total overall score; scoring is done for both sub-scores and summary scores.
Time Frame: Baseline, Month 12 (completion or termination)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 47 | 48
Score on a scale | 3.551 (8.351) | 2.846 (8.658)

18. Secondary Outcome: Area Under the Plasma Concentration of BAX 855 From Zero to Infinity (AUC0-inf)
Description: Area under the plasma concentration versus time curve from time 0 to infinity of BAX 855 were reported.
Time Frame: Pre-infusion, 15 - 30 minutes, 3, 8, 24, 48, 72 and 96 hours post-infusion
Population: Pharmacokinetic analysis set (PKAS) included all participants in the SAS that had at least one quantifiable post-dose FVIII activity level without major protocol deviations or events with potential to affect the PK analysis. Here "Number of participants analyzed" refer to number of participants evaluable for this outcome at specified time points.
Measure: Mean (Standard Deviation); unit: International units*hour per deciliter
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 54 | 57 | 5
International units*hour per deciliter | 2673 (877.3) | 2659 (1041) | 2214 (355.8)

19. Secondary Outcome: Incremental Recovery (IR) at Maximum Plasma Concentration (Cmax) of BAX 855
Description: IR at Cmax of BAX 855 were reported.
Time Frame: Pre-infusion, 15 - 30 minutes, 3, 8, 24, 48, 72 and 96 hours post-infusion
Population: PKAS included all participants in the SAS that had at least one quantifiable post-dose FVIII activity level without major protocol deviations or events with potential to affect the PK analysis. Here "Number of participants analyzed" refer to number of participants evaluable for this outcome at specified time points.
Measure: Mean (Standard Deviation); unit: (IU/dL) / (IU/kg)
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 57 | 58 | 5
(IU/dL) / (IU/kg) | 2.227 (0.5201) | 2.231 (0.5451) | 2.478 (0.2016)

20. Secondary Outcome: Plasma Half-life (T1/2) of BAX 855
Description: T1/2 of BAX 855 in plasma were reported.
Time Frame: Pre-infusion, 15 - 30 minutes, 3, 8, 24, 48, 72 and 96 hours post-infusion
Population: PKAS included all participants in the SAS that had at least one quantifiable post-dose FVIII activity level without major protocol deviations or events with potential to affect the PK analysis.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 57 | 58 | 5
hour (h) | 15.28 [8.77 to 31.9] | 14.66 [6.78 to 35.8] | 10.97 [8.67 to 12.5]

21. Secondary Outcome: Mean Residence Time (MRT) of BAX 855
Description: MRT of BAX 855 were reported.
Time Frame: Pre-infusion, 15 - 30 minutes, 3, 8, 24, 48, 72 and 96 hours post-infusion
Population: Pharmacokinetic analysis set (PKAS) included all participants in the SAS (participants enrolled who had at least 1 BAX 855 infusion) that had at least one quantifiable post-dose FVIII activity level without major protocol deviations or events with potential to affect the PK analysis.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 57 | 58 | 5
hour (h) | 22.77 [12.6 to 41.7] | 21.50 [10.1 to 52.5] | 16.18 [12.6 to 18.2]

22. Secondary Outcome: Maximum Plasma Concentration (Cmax) of BAX 855
Description: Cmax of BAX 855 were reported.
Time Frame: Pre-infusion, 15 - 30 minutes, 3, 8, 24, 48, 72 and 96 hours post-infusion
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: International units per deciliter(IU/dL)
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 54 | 57 | 5
International units per deciliter(IU/dL) | 132.54 (31.83) | 135.65 (33.10) | 149.18 (12.86)

23. Secondary Outcome: Time to Maximum Concentration of BAX 855 in Plasma (Tmax)
Description: Tmax of BAX 855 were reported.
Time Frame: Pre-infusion, 15 - 30 minutes, 3, 8, 24, 48, 72 and 96 hours post-infusion
Population: as for outcome 20
Measure: Median (Full Range); unit: hour (h)
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 57 | 58 | 5
hour (h) | 0.467 [0.30 to 3.08] | 0.475 [0.25 to 3.25] | 0.417 [0.38 to 0.53]

24. Secondary Outcome: Total Body Clearance (CL) of BAX 855
Description: Total body clearance of BAX 855 from blood by the kidney were reported.
Time Frame: Pre-infusion, 15 - 30 minutes, 3, 8, 24, 48, 72 and 96 hours post-infusion
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Deciliters per kilogram * hour (dL/kg*h)
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 57 | 58 | 5
Deciliters per kilogram * hour (dL/kg*h) | 0.02477 (0.009580) | 0.02624 (0.009333) | 0.02774 (0.004385)

25. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug was uniformly distributed to produce the desired blood concentration of a drug. Vss is the apparent volume of distribution at steadystate.
Time Frame: Pre-infusion, 15 - 30 minutes, 3, 8, 24, 48, 72 and 96 hours post-infusion
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Deciliters per kilogram (dL/kg)
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
Number analyzed (Participants) | 57 | 58 | 5
Deciliters per kilogram (dL/kg) | 0.5147 (0.1209) | 0.5158 (0.1062) | 149.18 (12.86)

26. Secondary Outcome: Incremental Recovery (IR) Over Time
Description: Incremental recovery was calculated by BAX 855 increment (IU/dL) / BAX 855 dose (IU/kg).
Time Frame: Baseline, Month 3, 6, 7.5, 9, 10.5, 12 (Completion or termination)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | BAX 855-Low Level | BAX 855-High Level
Number analyzed (Participants) | 57 | 58
IU/dL per IU/kg
  Baseline: number analyzed (Participants) | 53 | 54
  Baseline | 2.68 (0.513) | 2.70 (0.450)
  Month 3: number analyzed (Participants) | 56 | 54
  Month 3 | 2.68 (0.515) | 2.66 (0.459)
  Month 6: number analyzed (Participants) | 51 | 49
  Month 6 | 2.62 (0.585) | 2.76 (0.552)
  Month 7.5: number analyzed (Participants) | 13 | 11
  Month 7.5 | 2.53 (0.360) | 2.71 (0.545)
  Month 9: number analyzed (Participants) | 55 | 52
  Month 9 | 2.65 (0.511) | 2.68 (0.545)
  Month 10.5: number analyzed (Participants) | 12 | 5
  Month 10.5 | 2.61 (0.467) | 2.58 (0.584)
  Completion/ Termination: number analyzed (Participants) | 56 | 53
  Completion/ Termination | 2.71 (0.553) | 2.73 (0.689)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 12 months (completion or termination)
Arm/Group | BAX 855-Low Level | BAX 855-High Level | BAX 855-Non-randomized
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/58 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/57 | 5/58 | 0/6
Other Adverse Events (participants affected / at risk) | 25/57 | 25/58 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX 855-Low Level (N=57) | BAX 855-High Level (N=58) | BAX 855-Non-randomized (N=6)
Factor viii inhibition (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cerebellar haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX 855-Low Level (N=57) | BAX 855-High Level (N=58) | BAX 855-Non-randomized (N=6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (8) | 5 (6) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (11) | 12 (16) | 0 (0)
Headache (Nervous system disorders) | 5 (7) | 6 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (6):
  • Study Protocol: Protocol (2015-01-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT02585960/Prot_000.pdf
  • Study Protocol: Amendment 1 (2015-03-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT02585960/Prot_001.pdf
  • Study Protocol: Amendment 2 (2015-05-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT02585960/Prot_002.pdf
  • Study Protocol: Amendment 3 (2015-09-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT02585960/Prot_003.pdf
  • Study Protocol: Amendment 5 (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT02585960/Prot_004.pdf
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT02585960/SAP_005.pdf